CLINICAL TRIAL: NCT02663674
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial of Fluconazole as Early Empiric Treatment of Coccidioidomycosis Pneumonia (Valley Fever) in Adults Presenting With Community Acquired Pneumonia (CAP) in Endemic Areas (FLEET-Valley Fever)
Brief Title: Efficacy Study of Fluconazole to Treat Coccidioidomycosis Pneumonia (Valley Fever)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated due to lack of feasibility of study design.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-0053; HHSN272201300017I
Record Dates: First submitted 2016-01-15; First posted 2016-01-26 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-03

CONDITIONS: Coccidioidomycosis
Keywords: CAP; Coccidioidomycosis; Community Acquired Pneumonia; FLEET; Fluconazole; Parent Study of 16-0008; Pneumonia; Valley Fever
MeSH Terms: conditions — Coccidioidomycosis; Community-Acquired Pneumonia; Pneumonia | interventions — Fluconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Placebo Comparator): A single dose of Fluconazole placebo (2 capsules) administered orally once daily for 42 days starting on Day 1. N=500
  Interventions: Other: Placebo
- Group 2 (Experimental): 400 mg of Fluconazole (2 capsules of 200 mg) administered orally once daily for 42 days starting on Day 1. N=500
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Fluconazole — Fluconazole is a synthetic triazole antifungal agent. It will be supplied as 200 mg over encapsulated tablets. Each gelatin capsule will contain two-100 mg fluconazole tablets and microcrystalline cellulose for overfill.
  Arms: Group 2
Other: Placebo — Placebo will be supplied as matching gelatin capsules containing microcrystalline cellulose only. Capsules are the same size, weight, and color as capsules containing fluconazole tablets.
  Arms: Group 1

SUMMARY:
This is a Phase IV randomized, double-blinded, placebo-controlled study in 1000 individuals aged 18 years or older, with community acquired pneumonia (CAP) who meet all eligibility criteria in endemic regions. This study is designed to provide data on the effectiveness of early antifungal treatment (Fluconazole, 400 mg/day) for coccidioidomycosis pneumonia (also referred to as Valley Fever (VF) Pneumonia or acute onset valley fever) vs. placebo in subjects with coccidioidomycosis pneumonia. Patients who are prescribed antibacterials by their health care provider for acute CAP will be randomized to receive either placebo or 400 mg/day of fluconazole for 42 days. The primary objective is to assess the clinical response of early empiric antifungal therapy with fluconazole at Day 22 in subjects with coccidioidomycosis pneumonia and are compliant with the study intervention.

DETAILED DESCRIPTION:
This is a Phase IV randomized, double-blinded, placebo-controlled study in 1000 individuals, aged 18 years or older, with community acquired pneumonia (CAP) who meet all eligibility criteria in endemic regions. This study is designed to provide data on the effectiveness of early antifungal treatment (Fluconazole, 400 mg/day) for coccidioidomycosis pneumonia (also referred to as Valley Fever (VF) Pneumonia or acute onset valley fever) vs. placebo in subjects with coccidioidomycosis pneumonia. Patients who are prescribed antibacterials by their health care provider for acute CAP will be randomized to receive either placebo or 400 mg/day of fluconazole for 42 days. Blood work for serologic determination of coccidioidomycosis infection will be drawn at the time of randomization (Day 1), and again on Days, 22, 29, and 43. On Day 43, subjects will be informed of their treatment assignment and results of serologic testing from Days 1, 22 and 29. At Day 43, those subjects who did not meet the protocol defined case definition for CAP caused by acute coccidioidomycosis and who did not receive fluconazole will be dismissed from the study and referred to a health care provider with the results of their serology testing and their treatment assignment. All subjects who received fluconazole will be evaluated for safety follow up at Day 49. At Day 49, those subjects who did not meet the protocol defined case definition for CAP caused by acute coccidioidomycosis will be dismissed from the study and referred to a health care provider with the results of their serology testing and their treatment assignment. Subjects who did meet the protocol defined case definition for CAP caused by acute coccidioidomycosis infection will be referred to a healthcare provider with the results of their serology testing and their treatment assignment for further treatment as indicated and will be contacted by telephone on Days 90 and 180. The study duration will be approximately 72 months, and the subject participant duration will be from 42 days to approximately 6 months. The primary objective is to assess the clinical response of early empiric antifungal therapy with fluconazole at Day 22 in subjects with coccidioidomycosis pneumonia who are adherent to the study intervention. The secondary objectives are: 1) To assess the clinical response of early empiric antifungal therapy with fluconazole at Day 22 in subjects with coccidioidomycosis pneumonia regardless of adherence with the study intervention; 2) To assess the clinical response of early empiric antifungal therapy with fluconazole at Day 43 in subjects with coccidioidomycosis pneumonia regardless of adherence with the study intervention; 3) To compare the clinical response and its individual components over time, by treatment group, in subjects with coccidioidomycosis pneumonia; 4) To assess the impact of early empiric antifungal therapy with fluconazole on days lost from work or school and responses to the SF-12v2 and PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in subjects with coccidioidomycosis pneumonia; 5) To assess the effect of early empiric antifungal therapy with fluconazole through Day 43 in subjects with coccidioidomycosis pneumonia on all-cause mortality by treatment group; and 6) To assess whether early empiric antifungal therapy with fluconazole at Day 22 is non-inferior to placebo as defined by clinical response at Day 22 in all randomized subjects, regardless of coccidioidomycosis pneumonia status or adherence with study intervention, with baseline and follow-up FLEET-CAP scores.

ELIGIBILITY:
Inclusion Criteria:

1. Aged > / = 18 years and presenting for clinical care in coccidioidomycosis endemic areas.
2. Have a health care provider who has decided to treat community acquired pneumonia with antibacterials.
3. Be able to take and tolerate oral antibacterials/antifungals.
4. Able to understand the study and provide informed consent.
5. Willing and able to comply with study procedures and complete study visits.
6. Willing to allow access to medical records, and medical records are available to the study team.
7. The first dosage of study drug will be administered within 72 hours of presentation for care.
8. Able to swallow large pills.
9. Sexually active female subjects must be of non-childbearing potential* or, if of childbearing potential, must use a highly effective method of birth control**(captured on the appropriate data collection form).

   *Non-childbearing potential is defined as being post-menopausal for at least 18 months or surgically sterile via bilateral oophorectomy or hysterectomy.

   **Female subjects must avoid becoming pregnant by using one of the following acceptable methods of birth control for 30 days prior to study drug dosing and must be maintained for 30 days after last dose of study drug: i. Intrauterine contraceptive device; OR ii. Oral contraceptives; OR iii. Implanon, Nexplanon, DepoProvera, contraceptive skin patch or NuvaRing; OR iv. Tubal ligation; OR v. Exclusively same-sex relationships.
10. Non-pregnant female subjects of childbearing potential must have a negative pregnancy test within 24 hours prior to enrollment and at Visits 02 - 03.
11. Subjects receiving any of the drugs reported to have manageable drug interactions with fluconazole are allowed to be enrolled based on PI clinical judgment.

Exclusion Criteria:

1. Have recently received an experimental agent* or participating in or planning to participate in a study involving an experimental agent** while in the active drug administration phase of this study.

   *defined as within 30 days prior to enrollment in this study.

   **(e.g., vaccine, drug, biologic device, blood product, or medication).
2. Present clinical diagnosis of hospital acquired pneumonia (HAP).
3. Documented microbiologically- or serologically-confirmed past infection with coccidioidomycosis.
4. Clinical diagnosis of coccidioidal infection that is of sufficient certainty as to exclude the need for antibacterial therapy.
5. Have a history of systemic antibacterial treatment for this current CAP care episode occurring greater than 4 weeks prior to enrollment*.

   *Receipt of systemic antimicrobial therapy for indications other than respiratory tract infection is permitted.
6. Have a history of systemic antifungal treatment within the 4 weeks prior to enrollment.

   * A single dose of fluconazole (ex. treatment of vulvovaginal candidiasis) is acceptable and should not exclude subject from study.
7. Long term use* of high dose oral or parenteral glucocorticoids**; or high-dose inhaled steroids*** taken within the 4 weeks prior to enrollment.

   *defined as > 8 weeks of daily use.

   **high dose defined as prednisone > / = 20 mg total daily dose, or equivalent dose of other glucocorticoids.

   ***high dose defined as > 800 mcg/day of beclomethasone dipropionate or equivalent
8. Have confirmed or suspected immunosuppression as a result of an underlying illness [other than well controlled HIV infection], primary immunodeficiency, or treatment, or induction/maintenance use of immunosuppressive agents*.

   *including anti-neoplastic chemotherapy or cytotoxic radiation therapy for cancer, anti-TNF medications, or other immunomodulating agents.
9. History of a solid organ or bone marrow transplant.
10. Have poorly controlled HIV-infection or HIV-infection treated with Lopinavir, Tipranavir, Etravirine or Didanosine. Poorly controlled HIV is defined as HIV RNA > 50 copies/mm^3 (or greater than the lower limit of quantification [LLOQ] of the local HIV RNA assay if the LLOQ is > 50) in the 6 months prior to current care episode regardless of whether patient is on antiretroviral therapy or CD4 < 250 cell/mm^3.
11. Current diagnosis and/or treatment of active liver disease including abnormal baseline liver function tests as defined as: total bilirubin greater than or equal to 3.0 mg/dL AND either AST greater than or equal to 135 IU/L OR ALT greater than or equal to 150 IU/L.
12. On hemo or peritoneal dialysis or have a creatinine of > / = 2.0 mg/dL or estimated CrCl < /= 50 mL/min.
13. History of hypokalemia defined as less than 3.5 mEQ/L on more than one occasion during the 4 weeks prior to enrollment.
14. History of cardiovascular disease with increased risk for torsades de pointes as defined as: i. NYHA Heart Failure Criteria III or greater; OR ii. History of atrial or ventricular dysrhythmias; OR iii. History of structural heart disease (including previously repaired); OR iv.Personal or family history of congenital long QT syndrome.
15. A marked baseline prolongation of the QT/QTc interval defined as a QTc interval > 450 milliseconds (ms) for male subjects or > 470ms for female subjects with repeated demonstration*.

    *Subjects without a history of prolonged QTc and an abnormal baseline QTc interval should undergo repeat ECG assessment within screening period prior to randomization (72 hours) to confirm prolongation. If the repeat ECG QTc is within normal limits and less than the parameters above, the subject may be considered for enrollment.
16. Pregnant or lactating females.
17. History of azole intolerance or allergy.
18. Individuals for whom study participation would not be in their best interest, as determined by the clinical investigator.
19. Are taking medications that are contraindicated with concurrent use of fluconazole.
20. Positive point of care HIV test at Day 1 visit consistent with new HIV diagnosis.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-12-29 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Banner - University Medical Center Advanced Lung Disease Clinic - Phoenix, Phoenix, Arizona
  - St Josephs Hospital and Medical Center - Center for Liver Disease and Transplantation - Phoenix, Phoenix, Arizona
  - Mayo Clinic, Phoenix - Infectious Diseases, Phoenix, Arizona
  - Mayo Clinic, Scottsdale - Infectious Diseases, Scottsdale, Arizona
  - The University of Arizona - Banner University Medical Center Tucson Campus - Tucson, Tucson, Arizona
  - Kaiser Permanente Chester Avenue Medical Offices - Pulmonology, Bakersfield, California
  - Kern Medical Center - Medicine, Bakersfield, California
  - UCSF Fresno Center for Medical Education and Research - Clinical Research Center, Fresno, California
  - Kaiser Permanente Antelope Valley Medical Offices - Infectious Diseases, Lancaster, California

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between Feb 2016 and May 2018 at community locations in Coccidioides-endemic areas. Participants were adults presenting with community acquired pneumonia (CAP) whose health care provider had made the decision to treat with an antibacterial.
Groups:
- Fluconazole: Fluconazole was supplied as 200mg over encapsulated tablets. Each gelatin capsule contained two-100mg fluconazole tablets and microcrystalline cellulose for overfill. Fluconazole 400 mg (administered orally as two 200mg capsules) was to be taken once daily for a minimum of 42 days.
- Placebo: Placebo was supplied as matching gelatin capsules containing microcrystalline cellulose only. In order to maintain the blind, the gelatin capsules were the same size, weight, and color as the capsules containing fluconazole tablets. Placebo (administered orally as two matching placebo capsules) was to be taken once daily for a minimum of 42 days.
Period: Overall Study
Arm/Group | Fluconazole | Placebo
Started | 33 | 39
Completed | 26 | 29
Not Completed | 7 | 10
Not completed — Lost to Follow-up | 5 | 4
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Physician Decision | 1 | 1
Not completed — Other Event (Health Related) | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluconazole | Placebo | Total
Number analyzed (Participants) | 33 | 39 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 33 | 58
  >=65 years | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (16.1) | 49.5 (12.6) | 49.8 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 15 | 21 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 19 | 35
  Not Hispanic or Latino | 17 | 20 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 26 | 31 | 57
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 33 | 39 | 72
Positive for coccidioidomycosis pneumonia [Count of Participants; unit: Participants] — Participant diagnosed with CAP and meets one of the following criteria:
  1. Pos. for any 2 of IDTP, IDCF, EIA-IgM, EIA-IgG, between D1-D29, not necessarily from the same assay or same time point.
  2. Neg. for anti-Cocci antibody by ID (or EIA-IgG) at D1; seroconvert to pos. for anti-Cocci antibody by ID (or EIA-IgG) between D1-D29
  3. Neg. or indet. for anti-Cocci antibody by CF on D1; demonstrates a titer of >= 2 by CF between D1-D29
  4. Pos. for anti-Cocci antibody by CF on D1 and demonstrates a rise of >= 2-fold dilution in CF titer compared to baseline between D1-D29.
  Participants | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants Who Achieve a Clinical Response, Defined as at Least a 50% Reduction in Composite FLEET CAP Score From Baseline, in the Cocci-positive Per-protocol Population
Description: The Modified Scoring System for Evaluating Treatment Response in Early Coccidioidal Pneumonia (FLEET CAP) score is a clinical scoring system that allows a constellation of clinical symptoms to be quantified and scored over time: cough, fatigue, chest pain, dyspnea, sputum production, night sweats, fever and hypoxia. The recall period for symptom assessments was during the past week, with the exception of fever and hypoxia, which was measured on the day the FLEET CAP was administered. All symptoms are graded on a 0-3 severity scale, except for night sweats and hypoxia which are graded on a 0-2 severity scale, where 0 indicates the symptom is absent or normal. The range of total scores is from 0-22, where higher scores correspond to a worse outcome.
Time Frame: Visit 2 (Day 20-23)
Population: The cocci-positive per-protocol population includes randomized participants who met the case definition of cocci pneumonia, were adherent with the intervention and had coccidioidal serology data available at the Day 1 and 22 visits. To be considered adherent at the Day 22 visit, the participant needed to take >=80% of their expected capsules.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
Participants | 3 | 2

2. Secondary Outcome: The Proportion of Participants Who Achieve a Clinical Response, Defined as at Least a 50% Reduction in Composite FLEET CAP Score From Baseline, in the Cocci Positive Modified Intent-to-Treat Population
Description: as for outcome 1
Time Frame: Visit 2 (Day 20-23)
Population: Cocci Positive Modified Intent-to-Treat (mITT) population includes all randomized participants who meet the case definition of coccidioidomycosis pneumonia and took at least one dose of study medication. Note that it was not necessary for a participant to be adherent to study drug to be eligible for inclusion in the mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 3
Participants | 3 | 2

3. Secondary Outcome: The Proportion of Participants Who Achieve a Clinical Response, Defined as at Least a 50% Reduction in Composite FLEET CAP Score From Baseline, in the All Randomized mITT Population
Description: as for outcome 1
Time Frame: Visit 2 (Day 20-23)
Population: All Randomized Modified Intent-to-Treat (mITT) population - This efficacy analysis population includes all randomized participants who took at least one dose of study medication regardless of cocci-status. Note that it is not necessary for a participants to be adherent to study drug to be eligible for inclusion in the mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 27 | 35
Participants | 20 | 22

4. Secondary Outcome: The Proportion of Participants Who Achieve a Clinical Response, Defined as at Least a 50% Reduction in Composite FLEET CAP Score From Baseline, in All Randomized Participants Who Took at Least One Dose of Study Medication
Description: as for outcome 1
Time Frame: Visit 2 (Day 20-23)
Population: The population includes all participants who took at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 27 | 35
Participants | 20 | 22

5. Secondary Outcome: The Proportion of Participants Who Achieve a Clinical Response, Defined as at Least a 50% Reduction in Composite FLEET CAP Score From Baseline, in the Cocci Positive Modified Intent-to-Treat Population
Description: The Modified Scoring System for Evaluating Treatment Response in Early Coccidioidal Pneumonia (FLEET CAP) score is a clinical scoring system that allows a constellation of clinical symptoms to be quantified and scored over time: cough, fatigue, chest pain, dyspnea, sputum production, night sweats, fever and hypoxia. The recall period for symptom assessments was during the past week, with the exception of fever and hypoxia, which was measured on the day the FLEET CAP was administered. All symptoms are graded on a 0-3 severity scale, except for night sweats and hypoxia which are graded on a 0-2 severity scale, where 0 indicates the symptom is absent or normal. The range of total scores is from 0-22, where higher scores correspond to a worse outcome. Note that a participant who responds earlier before Day 43 does not need to achieve a clinical response at Day 43, as well.
Time Frame: Visit 2 - Visit 4 (Day 20-46)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
Participants | 4 | 2

6. Secondary Outcome: The Proportion of Participants Who Achieve a Clinical Response, Defined as at Least a 50% Reduction in Composite FLEET CAP Score From Baseline, in All Randomized Participants Who Took at Least One Dose of Study Medication
Description: as for outcome 5
Time Frame: Visit 2 - Visit 4 (Day 20-46)
Population: The population includes all participants who took at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 25 | 30
Participants | 25 | 28

7. Secondary Outcome: The Proportion of Participants Who Achieve a Clinical Response, Defined as at Least a 50% Reduction in Composite FLEET CAP Score From Baseline, in the All Randomized mITT Population
Description: as for outcome 5
Time Frame: Visit 2 - Visit 4 (Day 20-46)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 25 | 30
Participants | 25 | 28

8. Secondary Outcome: The Mean and Quartiles of the FLEET CAP Score and Each Component in the ITT Population
Description: as for outcome 1
Time Frame: Visit 2 (Day 20-23)
Population: The Intent-to-Treat (ITT) population includes all randomized participants.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 27 | 35
score on a scale
  Total FLEET CAP Score | 3.04 [1 to 5] | 3.49 [1 to 6]
  Cough | 0.85 [0 to 2] | 0.86 [0 to 1]
  Fatigue | 0.74 [0 to 1] | 0.74 [0 to 1]
  Chest Pain | 0.11 [0 to 0] | 0.31 [0 to 0]
  Dyspnea | 0.48 [0 to 1] | 0.60 [0 to 1]
  Sputum Production | 0.41 [0 to 1] | 0.40 [0 to 1]
  Night Sweats | 0.26 [0 to 0] | 0.37 [0 to 1]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0.19 [0 to 0] | 0.20 [0 to 0]

9. Secondary Outcome: The Median and Quartiles of the FLEET CAP Score and Each Component in the ITT Population
Description: as for outcome 1
Time Frame: Visit 2 (Day 20-23)
Population: The Intent-to-Treat (ITT) population includes all randomized participants.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 27 | 35
score on a scale
  Total FLEET CAP Score | 2.00 [1.00 to 5.00] | 2.00 [1.00 to 6.00]
  Cough | 1 [0 to 2] | 1 [0 to 1]
  Fatigue | 1 [0 to 1] | 0 [0 to 1]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0 [0 to 1] | 0 [0 to 1]
  Sputum Production | 0 [0 to 1] | 0 [0 to 1]
  Night Sweats | 0 [0 to 0] | 0 [0 to 1]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0 [0 to 0] | 0 [0 to 0]

10. Secondary Outcome: The Mean and Quartiles of the FLEET CAP Score and Each Component in the ITT Population
Description: as for outcome 1
Time Frame: Visit 3 (Day 27-30)
Population: The Intent-to-Treat (ITT) population includes all randomized participants.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 26 | 31
score on a scale
  Total FLEET CAP Score | 2.58 [0 to 4] | 1.97 [0 to 2]
  Cough | 0.73 [0 to 1] | 0.48 [0 to 1]
  Fatigue | 0.62 [0 to 1] | 0.42 [0 to 1]
  Chest Pain | 0.19 [0 to 0] | 0.13 [0 to 0]
  Dyspnea | 0.46 [0 to 1] | 0.42 [0 to 1]
  Sputum Production | 0.31 [0 to 0] | 0.16 [0 to 0]
  Night Sweats | 0.15 [0 to 0] | 0.19 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0.12 [0 to 0] | 0.16 [0 to 0]

11. Secondary Outcome: The Median and Quartiles of the FLEET CAP Score and Each Component in the ITT Population
Description: as for outcome 1
Time Frame: Visit 3 (Day 27-30)
Population: The Intent-to-Treat (ITT) population includes all randomized participants.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 26 | 31
score on a scale
  Total FLEET CAP Score | 2 [0 to 4] | 1 [0 to 2]
  Cough | 1 [0 to 1] | 0 [0 to 1]
  Fatigue | 0 [0 to 1] | 0 [0 to 1]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0 [0 to 1] | 0 [0 to 1]
  Sputum Production | 0 [0 to 0] | 0 [0 to 0]
  Night Sweats | 0 [0 to 0] | 0 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0 [0 to 0] | 0 [0 to 0]

12. Secondary Outcome: The Mean and Quartiles of the FLEET CAP Score and Each Component in the ITT Population
Description: as for outcome 1
Time Frame: Visit 4 (Day 42-46)
Population: The Intent-to-Treat (ITT) population includes all randomized participants.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 25 | 30
score on a scale
  Total FLEET CAP Score | 1.36 [0 to 2] | 1.5 [0 to 2]
  Cough | 0.44 [0 to 1] | 0.23 [0 to 0]
  Fatigue | 0.36 [0 to 1] | 0.37 [0 to 0]
  Chest Pain | 0.08 [0 to 0] | 0.17 [0 to 0]
  Dyspnea | 0.12 [0 to 0] | 0.30 [0 to 0]
  Sputum Production | 0.24 [0 to 0] | 0.13 [0 to 0]
  Night Sweats | 0.04 [0 to 0] | 0.10 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0.08 [0 to 0] | 0.20 [0 to 0]

13. Secondary Outcome: The Median and Quartiles of the FLEET CAP Score and Each Component in the ITT Population
Description: as for outcome 1
Time Frame: Visit 4 (Day 42-46)
Population: The Intent-to-Treat (ITT) population includes all randomized participants.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 25 | 30
score on a scale
  Total FLEET CAP Score | 1 [0 to 2] | 1 [0 to 2]
  Cough | 0 [0 to 1] | 0 [0 to 0]
  Fatigue | 0 [0 to 1] | 0 [0 to 0]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0 [0 to 0] | 0 [0 to 0]
  Sputum Production | 0 [0 to 0] | 0 [0 to 0]
  Night Sweats | 0 [0 to 0] | 0 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0 [0 to 0] | 0 [0 to 0]

14. Secondary Outcome: The Mean and Quartiles of the FLEET CAP Score and Each Component in the Cocci Positive Modified Intent-to-Treat (mITT) Population
Description: as for outcome 1
Time Frame: Visit 2 (Day 20-23)
Population: as for outcome 2
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 3
score on a scale
  Total FLEET CAP Score | 2.25 [1 to 3.5] | 3.67 [0 to 10]
  Cough | 0.5 [0 to 1] | 1 [0 to 2]
  Fatigue | 1.00 [0.5 to 1.5] | 1.00 [0 to 3]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0.5 [0 to 1] | 0.67 [0 to 2]
  Sputum Production | 0 [0 to 0] | 0.33 [0 to 1]
  Night Sweats | 0.25 [0 to 0.5] | 0.67 [0 to 2]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0 [0 to 0] | 0 [0 to 0]

15. Secondary Outcome: The Median and Quartiles of the FLEET CAP Score and Each Component in the Cocci Positive Modified Intent-to-Treat (mITT) Population
Description: as for outcome 1
Time Frame: Visit 2 (Day 20-23)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 3
score on a scale
  Total FLEET CAP Score | 1 [1 to 3.5] | 1 [0 to 10]
  Cough | 0 [0 to 1] | 1 [0 to 2]
  Fatigue | 1 [0.5 to 1.5] | 0 [0 to 3]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0 [0 to 1] | 0 [0 to 2]
  Sputum Production | 0 [0 to 0] | 0 [0 to 1]
  Night Sweats | 0 [0 to 0.5] | 0 [0 to 2]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0 [0 to 0] | 0 [0 to 0]

16. Secondary Outcome: The Mean and Quartiles of the FLEET CAP Score and Each Component in the Cocci Positive Modified Intent-to-Treat (mITT) Population
Description: as for outcome 1
Time Frame: Visit 3 (Day 27-30)
Population: as for outcome 2
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  Total FLEET CAP Score | 1.00 [0 to 2] | 0.5 [0 to 1]
  Cough | 0.5 [0 to 1] | 0 [0 to 0]
  Fatigue | 0.25 [0 to 0.5] | 0 [0 to 0]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0.25 [0 to 0.5] | 0.5 [0 to 1]
  Sputum Production | 0 [0 to 0] | 0 [0 to 0]
  Night Sweats | 0 [0 to 0] | 0 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0 [0 to 0] | 0 [0 to 0]

17. Secondary Outcome: The Median and Quartiles of the FLEET CAP Score and Each Component in the Cocci Positive Modified Intent-to-Treat (mITT) Population
Description: as for outcome 1
Time Frame: Visit 3 (Day 27-30)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  Total FLEET CAP Score | 0.5 [0 to 2] | 0.5 [0 to 1]
  Cough | 0.5 [0 to 1] | 0 [0 to 0]
  Fatigue | 0 [0 to 0.5] | 0 [0 to 0]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0 [0 to 0.5] | 0.5 [0 to 1]
  Sputum Production | 0 [0 to 0] | 0 [0 to 0]
  Night Sweats | 0 [0 to 0] | 0 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0 [0 to 0] | 0 [0 to 0]

18. Secondary Outcome: The Mean and Quartiles of the FLEET CAP Score and Each Component in the Cocci Positive Modified Intent-to-Treat (mITT) Population
Description: as for outcome 1
Time Frame: Visit 4 (Day 42-46)
Population: as for outcome 2
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  Total FLEET CAP Score | 0.75 [0 to 1.5] | 0 [0 to 0]
  Cough | 0.25 [0 to 0.5] | 0 [0 to 0]
  Fatigue | 0.25 [0 to 0.5] | 0 [0 to 0]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0 [0 to 0] | 0 [0 to 0]
  Sputum Production | 0 [0 to 0] | 0 [0 to 0]
  Night Sweats | 0 [0 to 0] | 0 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0.25 [0 to 0.5] | 0 [0 to 0]

19. Secondary Outcome: The Median and Quartiles of the FLEET CAP Score and Each Component in the Cocci Positive Modified Intent-to-Treat (mITT) Population
Description: as for outcome 1
Time Frame: Visit 4 (Day 42-46)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  Total FLEET CAP Score | 0 [0 to 1.5] | 0 [0 to 0]
  Cough | 0 [0 to 0.5] | 0 [0 to 0]
  Fatigue | 0 [0 to 0.5] | 0 [0 to 0]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0 [0 to 0] | 0 [0 to 0]
  Sputum Production | 0 [0 to 0] | 0 [0 to 0]
  Night Sweats | 0 [0 to 0] | 0 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0 [0 to 0.5] | 0 [0 to 0]

20. Secondary Outcome: The Mean and Quartiles of the FLEET CAP Score and Each Component in the All Randomized Modified Intent-to-Treat (mITT) Population
Description: as for outcome 1
Time Frame: Visit 2 (Day 20-23)
Population: as for outcome 3
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 27 | 35
score on a scale
  Total FLEET CAP Score | 3.04 [1 to 5] | 3.49 [1 to 6]
  Cough | 0.85 [0 to 2] | 0.86 [0 to 1]
  Fatigue | 0.74 [0 to 1] | 0.74 [0 to 1]
  Chest Pain | 0.11 [0 to 0] | 0.31 [0 to 0]
  Dyspnea | 0.48 [0 to 1] | 0.6 [0 to 1]
  Sputum Production | 0.41 [0 to 1] | 0.40 [0 to 1]
  Night Sweats | 0.26 [0 to 0] | 0.37 [0 to 1]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0.19 [0 to 0] | 0.20 [0 to 0]

21. Secondary Outcome: The Median and Quartiles of the FLEET CAP Score and Each Component in the All Randomized Modified Intent-to-Treat (mITT) Population
Description: as for outcome 1
Time Frame: Visit 2 (Day 20-23)
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 27 | 35
score on a scale
  Total FLEET CAP Score | 2 [1 to 5] | 2 [1 to 6]
  Cough | 1 [0 to 2] | 1 [0 to 1]
  Fatigue | 1 [0 to 1] | 0 [0 to 1]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0 [0 to 1] | 0 [0 to 1]
  Sputum Production | 0 [0 to 1] | 0 [0 to 1]
  Night Sweats | 0 [0 to 0] | 0 [0 to 1]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0 [0 to 0] | 0 [0 to 0]

22. Secondary Outcome: The Mean and Quartiles of the FLEET CAP Score and Each Component in the All Randomized Modified Intent-to-Treat (mITT) Population
Description: as for outcome 1
Time Frame: Visit 3 (Day 27-30)
Population: as for outcome 3
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 26 | 31
score on a scale
  Total FLEET CAP Score | 2.58 [0 to 4] | 1.97 [0 to 2]
  Cough | 0.73 [0 to 1] | 0.48 [0 to 1]
  Fatigue | 0.62 [0 to 1] | 0.42 [0 to 1]
  Chest Pain | 0.19 [0 to 0] | 0.13 [0 to 0]
  Dyspnea | 0.46 [0 to 1] | 0.42 [0 to 1]
  Sputum Production | 0.31 [0 to 0] | 0.16 [0 to 0]
  Night Sweats | 0.15 [0 to 0] | 0.19 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0.12 [0 to 0] | 0.16 [0 to 0]

23. Secondary Outcome: The Median and Quartiles of the FLEET CAP Score and Each Component in the All Randomized Modified Intent-to-Treat (mITT) Population
Description: as for outcome 1
Time Frame: Visit 3 (Day 27-30)
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 26 | 31
score on a scale
  Total FLEET CAP Score | 2 [0 to 4] | 1 [0 to 2]
  Cough | 1 [0 to 1] | 0 [0 to 1]
  Fatigue | 0 [0 to 1] | 0 [0 to 1]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0 [0 to 1] | 0 [0 to 1]
  Sputum Production | 0 [0 to 0] | 0 [0 to 0]
  Night Sweats | 0 [0 to 0] | 0 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0 [0 to 0] | 0 [0 to 0]

24. Secondary Outcome: The Mean and Quartiles of the FLEET CAP Score and Each Component in the All Randomized Modified Intent-to-Treat (mITT) Population
Description: as for outcome 1
Time Frame: Visit 4 (Day 42-46)
Population: as for outcome 3
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 25 | 30
score on a scale
  Total FLEET CAP Score | 1.36 [0 to 2] | 1.5 [0 to 2]
  Cough | 0.44 [0 to 1] | 0.23 [0 to 0]
  Fatigue | 0.36 [0 to 1] | 0.37 [0 to 0]
  Chest Pain | 0.08 [0 to 0] | 0.17 [0 to 0]
  Dyspnea | 0.12 [0 to 0] | 0.30 [0 to 0]
  Sputum Production | 0.24 [0 to 0] | 0.13 [0 to 0]
  Night Sweats | 0.04 [0 to 0] | 0.10 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0.08 [0 to 0] | 0.20 [0 to 0]

25. Secondary Outcome: The Median and Quartiles of the FLEET CAP Score and Each Component in the All Randomized Modified Intent-to-Treat (mITT) Population
Description: as for outcome 1
Time Frame: Visit 4 (Day 42-46)
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 25 | 30
score on a scale
  Total FLEET CAP Score | 1 [0 to 2] | 1 [0 to 2]
  Cough | 0 [0 to 1] | 0 [0 to 0]
  Fatigue | 0 [0 to 1] | 0 [0 to 0]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0 [0 to 0] | 0 [0 to 0]
  Sputum Production | 0 [0 to 0] | 0 [0 to 0]
  Night Sweats | 0 [0 to 0] | 0 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0 [0 to 0] | 0 [0 to 0]

26. Secondary Outcome: The Mean and Quartiles of the FLEET CAP Score and Each Component in the Cocci Positive Per-Protocol (PP) Population
Description: as for outcome 1
Time Frame: Visit 2 (Day 20-23)
Population: The cocci-positive per-protocol population includes randomized participants who met the case definition of cocci pneumonia, were adherent with the intervention and had coccidioidal serology data available at the Day 1 and 22 visits. To be considered adherent at the Day 22 visit, the participant needed to take >=80% of their expected pills.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  Total FLEET CAP Score | 2.25 [1 to 3.5] | 0.5 [0 to 1]
  Cough | 0.5 [0 to 1] | 0.5 [0 to 1]
  Fatigue | 1.00 [0.5 to 1.5] | 0 [0 to 0]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0.5 [0 to 1] | 0 [0 to 0]
  Sputum Production | 0 [0 to 0] | 0 [0 to 0]
  Night Sweats | 0.25 [0 to 0.5] | 0 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0 [0 to 0] | 0 [0 to 0]

27. Secondary Outcome: The Median and Quartiles of the FLEET CAP Score and Each Component in the Cocci Positive Per-Protocol (PP) Population
Description: as for outcome 1
Time Frame: Visit 2 (Day 20-23)
Population: as for outcome 26
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  Total FLEET CAP Score | 1 [1 to 3.5] | 0.5 [0 to 1]
  Cough | 0 [0 to 1] | 0.5 [0 to 1]
  Fatigue | 1 [0.5 to 1.5] | 0 [0 to 0]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0 [0 to 1] | 0 [0 to 0]
  Sputum Production | 0 [0 to 0] | 0 [0 to 0]
  Night Sweats | 0 [0 to 0.5] | 0 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0 [0 to 0] | 0 [0 to 0]

28. Secondary Outcome: The Mean and Quartiles of the FLEET CAP Score and Each Component in the Cocci Positive Per-Protocol (PP) Population
Description: as for outcome 1
Time Frame: Visit 3 (Day 27-30)
Population: as for outcome 26
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  Total FLEET CAP Score | 1.00 [0 to 2] | 0.5 [0 to 1]
  Cough | 0.5 [0 to 1] | 0 [0 to 0]
  Fatigue | 0.25 [0 to 0.5] | 0 [0 to 0]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0.25 [0 to 0.5] | 0.5 [0 to 1]
  Sputum Production | 0 [0 to 0] | 0 [0 to 0]
  Night Sweats | 0 [0 to 0] | 0 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0 [0 to 0] | 0 [0 to 0]

29. Secondary Outcome: The Median and Quartiles of the FLEET CAP Score and Each Component in the Cocci Positive Per-Protocol (PP) Population
Description: as for outcome 1
Time Frame: Visit 3 (Day 27-30)
Population: as for outcome 26
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  Total FLEET CAP Score | 0.5 [0 to 2] | 0.5 [0 to 1]
  Cough | 0.5 [0 to 1] | 0 [0 to 0]
  Fatigue | 0 [0 to 0.5] | 0 [0 to 0]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0 [0 to 0.5] | 0.5 [0 to 1]
  Sputum Production | 0 [0 to 0] | 0 [0 to 0]
  Night Sweats | 0 [0 to 0] | 0 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0 [0 to 0] | 0 [0 to 0]

30. Secondary Outcome: The Mean and Quartiles of the FLEET CAP Score and Each Component in the Cocci Positive Per-Protocol (PP) Population
Description: as for outcome 1
Time Frame: Visit 4 (Day 42-46)
Population: as for outcome 26
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  Total FLEET CAP Score | 0.75 [0 to 1.5] | 0 [0 to 0]
  Cough | 0.25 [0 to 0.5] | 0 [0 to 0]
  Fatigue | 0.25 [0 to 0.5] | 0 [0 to 0]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0 [0 to 0] | 0 [0 to 0]
  Sputum Production | 0 [0 to 0] | 0 [0 to 0]
  Night Sweats | 0 [0 to 0] | 0 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0.25 [0 to 0.5] | 0 [0 to 0]

31. Secondary Outcome: The Median and Quartiles of the FLEET CAP Score and Each Component in the Cocci Positive Per-Protocol (PP) Population
Description: as for outcome 1
Time Frame: Visit 4 (Day 42-46)
Population: as for outcome 26
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  Total FLEET CAP Score | 0 [0 to 1.5] | 0 [0 to 0]
  Cough | 0 [0 to 0.5] | 0 [0 to 0]
  Fatigue | 0 [0 to 0.5] | 0 [0 to 0]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0 [0 to 0] | 0 [0 to 0]
  Sputum Production | 0 [0 to 0] | 0 [0 to 0]
  Night Sweats | 0 [0 to 0] | 0 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0 [0 to 0.5] | 0 [0 to 0]

32. Secondary Outcome: The Mean and Quartiles of the FLEET CAP Score and Each Component in the All Randomized Per-Protocol (PP) Population
Description: as for outcome 1
Time Frame: Visit 2 (Day 20-23)
Population: The All Randomized Per-Protocol (PP) population includes randomized participants who were compliant with the intervention administration regardless of cocci-status and have coccidioidal serology data available at the Day 1 and 22 visits.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 25 | 29
score on a scale
  Total FLEET CAP Score | 2.64 [1 to 4] | 3.72 [1 to 6]
  Cough | 0.80 [0 to 1] | 0.97 [0 to 1]
  Fatigue | 0.72 [0 to 1] | 0.76 [0 to 1]
  Chest Pain | 0.08 [0 to 0] | 0.34 [0 to 0]
  Dyspnea | 0.40 [0 to 1] | 0.66 [0 to 1]
  Sputum Production | 0.32 [0 to 1] | 0.45 [0 to 1]
  Night Sweats | 0.16 [0 to 0] | 0.38 [0 to 1]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0.16 [0 to 0] | 0.17 [0 to 0]

33. Secondary Outcome: The Median and Quartiles of the FLEET CAP Score and Each Component in the All Randomized Per-Protocol (PP) Population
Description: as for outcome 1
Time Frame: Visit 2 (Day 20-23)
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 25 | 29
score on a scale
  Total FLEET CAP Score | 2 [1 to 4] | 3 [1 to 6]
  Cough | 1 [0 to 1] | 1 [0 to 1]
  Fatigue | 1 [0 to 1] | 0 [0 to 1]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0 [0 to 1] | 0 [0 to 1]
  Sputum Production | 0 [0 to 1] | 0 [0 to 1]
  Night Sweats | 0 [0 to 0] | 0 [0 to 1]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0 [0 to 0] | 0 [0 to 0]

34. Secondary Outcome: The Mean and Quartiles of the FLEET CAP Score and Each Component in the All Randomized Per-Protocol (PP) Population
Description: as for outcome 1
Time Frame: Visit 3 (Day 27-30)
Population: as for outcome 32
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 24 | 25
score on a scale
  Total FLEET CAP Score | 2.42 [0 to 3.5] | 1.96 [0 to 2]
  Cough | 0.71 [0 to 1] | 0.48 [0 to 1]
  Fatigue | 0.63 [0 to 1] | 0.44 [0 to 1]
  Chest Pain | 0.17 [0 to 0] | 0.12 [0 to 0]
  Dyspnea | 0.42 [0 to 1] | 0.44 [0 to 1]
  Sputum Production | 0.33 [0 to .5] | 0.16 [0 to 0]
  Night Sweats | 0.08 [0 to 0] | 0.20 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0.08 [0 to 0] | 0.12 [0 to 0]

35. Secondary Outcome: The Median and Quartiles of the FLEET CAP Score and Each Component in the All Randomized Per-Protocol (PP) Population
Description: as for outcome 1
Time Frame: Visit 3 (Day 27-30)
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 24 | 25
score on a scale
  Total FLEET CAP Score | 2 [0 to 3.5] | 1 [0 to 2]
  Cough | 1 [0 to 1] | 0 [0 to 1]
  Fatigue | 0 [0 to 1] | 0 [0 to 1]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0 [0 to 1] | 0 [0 to 1]
  Sputum Production | 0 [0 to 0.5] | 0 [0 to 0]
  Night Sweats | 0 [0 to 0] | 0 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0 [0 to 0] | 0 [0 to 0]

36. Secondary Outcome: The Mean and Quartiles of the FLEET CAP Score and Each Component in the All Randomized Per-Protocol (PP) Population
Description: as for outcome 1
Time Frame: Visit 4 (Day 42-46)
Population: as for outcome 32
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 23 | 24
score on a scale
  Total FLEET CAP Score | 1.09 [0 to 2] | 1.25 [0 to 2]
  Cough | 0.35 [0 to 1] | 0.21 [0 to 0]
  Fatigue | 0.35 [0 to 1] | 0.38 [0 to 0]
  Chest Pain | 0.04 [0 to 0] | 0.13 [0 to 0]
  Dyspnea | 0.09 [0 to 0] | 0.21 [0 to 0]
  Sputum Production | 0.13 [0 to 0] | 0.08 [0 to 0]
  Night Sweats | 0.04 [0 to 0] | 0.08 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0.09 [0 to 0] | 0.17 [0 to 0]

37. Secondary Outcome: The Median and Quartiles of the FLEET CAP Score and Each Component in the All Randomized Per-Protocol (PP) Population
Description: as for outcome 1
Time Frame: Visit 4 (Day 42-46)
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 23 | 24
score on a scale
  Total FLEET CAP Score | 0 [0 to 2] | 0.5 [0 to 2]
  Cough | 0 [0 to 1] | 0 [0 to 0]
  Fatigue | 0 [0 to 1] | 0 [0 to 0]
  Chest Pain | 0 [0 to 0] | 0 [0 to 0]
  Dyspnea | 0 [0 to 0] | 0 [0 to 0]
  Sputum Production | 0 [0 to 0] | 0 [0 to 0]
  Night Sweats | 0 [0 to 0] | 0 [0 to 0]
  Fever | 0 [0 to 0] | 0 [0 to 0]
  Hypoxia | 0 [0 to 0] | 0 [0 to 0]

38. Secondary Outcome: Number of the Days of School or Work Missed Due to Illness in the ITT Population
Description: Number of the days of school or work missed due to illness by participant self-report
Time Frame: Visit 1 (Day 1) through Visit 4 (Day 42-46)
Population: The Intent-to-Treat (ITT) population includes all randomized participants.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 19 | 23
days | 0 (0) | 1.5 (5.2)

39. Secondary Outcome: Number of the Days of School or Work Missed Due to Illness in the Cocci Positive mITT Population
Description: Number of the days of school or work missed due to illness by participant self-report
Time Frame: Visit 1 (Day 1) through Visit 4 (Day 42-46)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 2 | 0
days | 0 (0) |

40. Secondary Outcome: Number of the Days of School or Work Missed Due to Illness in the All Randomized PP Population
Description: Number of the days of school or work missed due to illness by participant self-report
Time Frame: Visit 1 (Day 1) through Visit 4 (Day 42-46)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 18 | 17
days | 0 (0) | 0.6 (1.8)

41. Secondary Outcome: Number of the Days of School or Work Missed Due to Illness in the Cocci Positive PP Population
Description: Number of the days of school or work missed due to illness by participant self-report
Time Frame: Visit 1 (Day 1) through Visit 4 (Day 42-46)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 2 | 0
days | 0 (0) |

42. Secondary Outcome: Number of the Days of School or Work Missed Due to Illness in the All Randomized mITT Population
Description: Number of the days of school or work missed due to illness by participant self-report
Time Frame: Visit 1 (Day 1) through Visit 4 (Day 42-46)
Population: All Randomized Modified Intent-to-Treat (mITT) population - This efficacy analysis population includes all randomized participants who took at least one dose of study medication regardless of cocci-status. Note that it is not necessary for a participant to be adherent to study drug to be eligible for inclusion in the mITT population.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 19 | 23
days | 0 (0) | 1.5 (5.2)

43. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the ITT Population
Description: The PROMIS Ability to Participate in Social Roles and Activities - Short Form 4a uses 4 questions to measure the participant's ability to participate in social roles and activities in the context of family, friends, leisure, and work. Four individual items are answered as "Never", "Rarely", "Sometimes", "Usually", or "Always" with an "Always" response indicating the most trouble participating in social roles and activities.
Time Frame: Visit 2 (Day 20-23)
Population: The Intent-to-Treat (ITT) population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 27 | 35
Participants
  Trouble doing regular leisure activities w others: Never | 1 | 3
  Trouble doing regular leisure activities w others: Rarely | 1 | 4
  Trouble doing regular leisure activities w others: Sometimes | 7 | 8
  Trouble doing regular leisure activities w others: Usually | 3 | 7
  Trouble doing regular leisure activities w others: Always | 15 | 13
  Trouble doing family activities I want to do: Never | 0 | 3
  Trouble doing family activities I want to do: Rarely | 3 | 4
  Trouble doing family activities I want to do: Sometimes | 4 | 7
  Trouble doing family activities I want to do: Usually | 5 | 6
  Trouble doing family activities I want to do: Always | 15 | 15
  Trouble doing usual work (incl work at home): Never | 0 | 3
  Trouble doing usual work (incl work at home): Rarely | 5 | 4
  Trouble doing usual work (incl work at home): Sometimes | 7 | 9
  Trouble doing usual work (incl work at home): Usually | 4 | 6
  Trouble doing usual work (incl work at home): Always | 11 | 13
  Trouble doing activities with friends I want to do: Never | 1 | 4
  Trouble doing activities with friends I want to do: Rarely | 3 | 2
  Trouble doing activities with friends I want to do: Sometimes | 5 | 10
  Trouble doing activities with friends I want to do: Usually | 4 | 7
  Trouble doing activities with friends I want to do: Always | 14 | 12

44. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the ITT Population
Description: as for outcome 43
Time Frame: Visit 3 (Day 27-30)
Population: The Intent-to-Treat (ITT) population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 26 | 31
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 3 | 1
  Trouble doing regular leisure activities w others: Sometimes | 6 | 8
  Trouble doing regular leisure activities w others: Usually | 4 | 13
  Trouble doing regular leisure activities w others: Always | 13 | 9
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 2 | 1
  Trouble doing family activities I want to do: Sometimes | 6 | 11
  Trouble doing family activities I want to do: Usually | 4 | 10
  Trouble doing family activities I want to do: Always | 14 | 9
  Trouble doing usual work (incl work at home): Never | 0 | 0
  Trouble doing usual work (incl work at home): Rarely | 4 | 3
  Trouble doing usual work (incl work at home): Sometimes | 5 | 10
  Trouble doing usual work (incl work at home): Usually | 4 | 10
  Trouble doing usual work (incl work at home): Always | 13 | 8
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 2 | 3
  Trouble doing activities with friends I want to do: Sometimes | 6 | 7
  Trouble doing activities with friends I want to do: Usually | 5 | 10
  Trouble doing activities with friends I want to do: Always | 13 | 11

45. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the ITT Population
Description: as for outcome 43
Time Frame: Visit 4 (Day 42-46)
Population: The Intent-to-Treat (ITT) population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 25 | 30
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 1 | 4
  Trouble doing regular leisure activities w others: Sometimes | 6 | 6
  Trouble doing regular leisure activities w others: Usually | 4 | 8
  Trouble doing regular leisure activities w others: Always | 14 | 12
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 2 | 4
  Trouble doing family activities I want to do: Sometimes | 5 | 5
  Trouble doing family activities I want to do: Usually | 2 | 6
  Trouble doing family activities I want to do: Always | 16 | 15
  Trouble doing usual work (incl work at home): Never | 1 | 0
  Trouble doing usual work (incl work at home): Rarely | 1 | 4
  Trouble doing usual work (incl work at home): Sometimes | 5 | 4
  Trouble doing usual work (incl work at home): Usually | 4 | 11
  Trouble doing usual work (incl work at home): Always | 14 | 11
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 2 | 5
  Trouble doing activities with friends I want to do: Sometimes | 5 | 5
  Trouble doing activities with friends I want to do: Usually | 4 | 4
  Trouble doing activities with friends I want to do: Always | 14 | 16

46. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the ITT Population
Description: as for outcome 43
Time Frame: Visit 6 (Day 83-97)
Population: The Intent-to-Treat (ITT) population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 0 | 0
  Trouble doing regular leisure activities w others: Sometimes | 1 | 0
  Trouble doing regular leisure activities w others: Usually | 0 | 0
  Trouble doing regular leisure activities w others: Always | 3 | 1
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 0 | 0
  Trouble doing family activities I want to do: Sometimes | 1 | 0
  Trouble doing family activities I want to do: Usually | 0 | 0
  Trouble doing family activities I want to do: Always | 3 | 1
  Trouble doing usual work (incl work at home): Never | 1 | 0
  Trouble doing usual work (incl work at home): Rarely | 0 | 0
  Trouble doing usual work (incl work at home): Sometimes | 0 | 0
  Trouble doing usual work (incl work at home): Usually | 0 | 0
  Trouble doing usual work (incl work at home): Always | 3 | 1
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 0 | 0
  Trouble doing activities with friends I want to do: Sometimes | 1 | 0
  Trouble doing activities with friends I want to do: Usually | 0 | 0
  Trouble doing activities with friends I want to do: Always | 3 | 1

47. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the ITT Population
Description: as for outcome 43
Time Frame: Visit 7 (Day 173-187)
Population: The Intent-to-Treat (ITT) population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 1 | 0
  Trouble doing regular leisure activities w others: Sometimes | 0 | 0
  Trouble doing regular leisure activities w others: Usually | 0 | 0
  Trouble doing regular leisure activities w others: Always | 3 | 1
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 0 | 0
  Trouble doing family activities I want to do: Sometimes | 0 | 0
  Trouble doing family activities I want to do: Usually | 1 | 0
  Trouble doing family activities I want to do: Always | 3 | 1
  Trouble doing usual work (incl work at home): Never | 0 | 0
  Trouble doing usual work (incl work at home): Rarely | 0 | 0
  Trouble doing usual work (incl work at home): Sometimes | 1 | 0
  Trouble doing usual work (incl work at home): Usually | 0 | 0
  Trouble doing usual work (incl work at home): Always | 3 | 1
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 1 | 0
  Trouble doing activities with friends I want to do: Sometimes | 0 | 0
  Trouble doing activities with friends I want to do: Usually | 0 | 0
  Trouble doing activities with friends I want to do: Always | 3 | 1

48. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the Cocci Positive Per Protocol Population
Description: as for outcome 43
Time Frame: Visit 2 (Day 20-23)
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 0 | 0
  Trouble doing regular leisure activities w others: Sometimes | 1 | 1
  Trouble doing regular leisure activities w others: Usually | 0 | 0
  Trouble doing regular leisure activities w others: Always | 3 | 1
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 0 | 0
  Trouble doing family activities I want to do: Sometimes | 1 | 0
  Trouble doing family activities I want to do: Usually | 0 | 1
  Trouble doing family activities I want to do: Always | 3 | 1
  Trouble doing usual work (incl work at home): Never | 0 | 0
  Trouble doing usual work (incl work at home): Rarely | 1 | 0
  Trouble doing usual work (incl work at home): Sometimes | 0 | 1
  Trouble doing usual work (incl work at home): Usually | 1 | 0
  Trouble doing usual work (incl work at home): Always | 2 | 1
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 0 | 0
  Trouble doing activities with friends I want to do: Sometimes | 1 | 1
  Trouble doing activities with friends I want to do: Usually | 0 | 0
  Trouble doing activities with friends I want to do: Always | 3 | 1

49. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the Cocci Positive Per Protocol Population
Description: as for outcome 43
Time Frame: Visit 3 (Day 27-30)
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 0 | 0
  Trouble doing regular leisure activities w others: Sometimes | 1 | 0
  Trouble doing regular leisure activities w others: Usually | 1 | 1
  Trouble doing regular leisure activities w others: Always | 2 | 1
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 1 | 0
  Trouble doing family activities I want to do: Sometimes | 0 | 0
  Trouble doing family activities I want to do: Usually | 1 | 1
  Trouble doing family activities I want to do: Always | 2 | 1
  Trouble doing usual work (incl work at home): Never | 0 | 0
  Trouble doing usual work (incl work at home): Rarely | 1 | 0
  Trouble doing usual work (incl work at home): Sometimes | 0 | 0
  Trouble doing usual work (incl work at home): Usually | 1 | 1
  Trouble doing usual work (incl work at home): Always | 2 | 1
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 0 | 0
  Trouble doing activities with friends I want to do: Sometimes | 1 | 0
  Trouble doing activities with friends I want to do: Usually | 1 | 1
  Trouble doing activities with friends I want to do: Always | 2 | 1

50. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the Cocci Positive Per Protocol Population
Description: as for outcome 43
Time Frame: Visit 4 (Day 42-46)
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 0 | 0
  Trouble doing regular leisure activities w others: Sometimes | 1 | 0
  Trouble doing regular leisure activities w others: Usually | 0 | 0
  Trouble doing regular leisure activities w others: Always | 3 | 2
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 0 | 0
  Trouble doing family activities I want to do: Sometimes | 1 | 0
  Trouble doing family activities I want to do: Usually | 0 | 0
  Trouble doing family activities I want to do: Always | 3 | 2
  Trouble doing usual work (incl work at home): Never | 0 | 0
  Trouble doing usual work (incl work at home): Rarely | 1 | 0
  Trouble doing usual work (incl work at home): Sometimes | 0 | 0
  Trouble doing usual work (incl work at home): Usually | 0 | 1
  Trouble doing usual work (incl work at home): Always | 3 | 1
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 0 | 0
  Trouble doing activities with friends I want to do: Sometimes | 1 | 0
  Trouble doing activities with friends I want to do: Usually | 0 | 0
  Trouble doing activities with friends I want to do: Always | 3 | 2

51. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the Cocci Positive Per Protocol Population
Description: as for outcome 43
Time Frame: Visit 6 (Day 83-97)
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 0 | 0
  Trouble doing regular leisure activities w others: Sometimes | 1 | 0
  Trouble doing regular leisure activities w others: Usually | 0 | 0
  Trouble doing regular leisure activities w others: Always | 3 | 1
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 0 | 0
  Trouble doing family activities I want to do: Sometimes | 1 | 0
  Trouble doing family activities I want to do: Usually | 0 | 0
  Trouble doing family activities I want to do: Always | 3 | 1
  Trouble doing usual work (incl work at home): Never | 1 | 0
  Trouble doing usual work (incl work at home): Rarely | 0 | 0
  Trouble doing usual work (incl work at home): Sometimes | 0 | 0
  Trouble doing usual work (incl work at home): Usually | 0 | 0
  Trouble doing usual work (incl work at home): Always | 3 | 1
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 0 | 0
  Trouble doing activities with friends I want to do: Sometimes | 1 | 0
  Trouble doing activities with friends I want to do: Usually | 0 | 0
  Trouble doing activities with friends I want to do: Always | 3 | 1

52. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the Cocci Positive Per Protocol Population
Description: as for outcome 43
Time Frame: Visit 7 (Day 173-187)
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 1 | 0
  Trouble doing regular leisure activities w others: Sometimes | 0 | 0
  Trouble doing regular leisure activities w others: Usually | 0 | 0
  Trouble doing regular leisure activities w others: Always | 3 | 1
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 0 | 0
  Trouble doing family activities I want to do: Sometimes | 0 | 0
  Trouble doing family activities I want to do: Usually | 1 | 0
  Trouble doing family activities I want to do: Always | 3 | 1
  Trouble doing usual work (incl work at home): Never | 0 | 0
  Trouble doing usual work (incl work at home): Rarely | 0 | 0
  Trouble doing usual work (incl work at home): Sometimes | 1 | 0
  Trouble doing usual work (incl work at home): Usually | 0 | 0
  Trouble doing usual work (incl work at home): Always | 3 | 1
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 1 | 0
  Trouble doing activities with friends I want to do: Sometimes | 0 | 0
  Trouble doing activities with friends I want to do: Usually | 0 | 0
  Trouble doing activities with friends I want to do: Always | 3 | 1

53. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the Cocci Positive mITT Population
Description: as for outcome 43
Time Frame: Visit 2 (Day 20-23)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 3
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 1
  Trouble doing regular leisure activities w others: Rarely | 0 | 0
  Trouble doing regular leisure activities w others: Sometimes | 1 | 1
  Trouble doing regular leisure activities w others: Usually | 0 | 0
  Trouble doing regular leisure activities w others: Always | 3 | 1
  Trouble doing family activities I want to do: Never | 0 | 1
  Trouble doing family activities I want to do: Rarely | 0 | 0
  Trouble doing family activities I want to do: Sometimes | 1 | 0
  Trouble doing family activities I want to do: Usually | 0 | 1
  Trouble doing family activities I want to do: Always | 3 | 1
  Trouble doing usual work (incl work at home): Never | 0 | 1
  Trouble doing usual work (incl work at home): Rarely | 1 | 0
  Trouble doing usual work (incl work at home): Sometimes | 0 | 1
  Trouble doing usual work (incl work at home): Usually | 1 | 0
  Trouble doing usual work (incl work at home): Always | 2 | 1
  Trouble doing activities with friends I want to do: Never | 0 | 1
  Trouble doing activities with friends I want to do: Rarely | 0 | 0
  Trouble doing activities with friends I want to do: Sometimes | 1 | 1
  Trouble doing activities with friends I want to do: Usually | 0 | 0
  Trouble doing activities with friends I want to do: Always | 3 | 1

54. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the Cocci Positive mITT Population
Description: as for outcome 43
Time Frame: Visit 3 (Day 27-30)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 0 | 0
  Trouble doing regular leisure activities w others: Sometimes | 1 | 0
  Trouble doing regular leisure activities w others: Usually | 1 | 1
  Trouble doing regular leisure activities w others: Always | 2 | 1
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 1 | 0
  Trouble doing family activities I want to do: Sometimes | 0 | 0
  Trouble doing family activities I want to do: Usually | 1 | 1
  Trouble doing family activities I want to do: Always | 2 | 1
  Trouble doing usual work (incl work at home): Never | 0 | 0
  Trouble doing usual work (incl work at home): Rarely | 1 | 0
  Trouble doing usual work (incl work at home): Sometimes | 0 | 0
  Trouble doing usual work (incl work at home): Usually | 1 | 1
  Trouble doing usual work (incl work at home): Always | 2 | 1
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 0 | 0
  Trouble doing activities with friends I want to do: Sometimes | 1 | 0
  Trouble doing activities with friends I want to do: Usually | 1 | 1
  Trouble doing activities with friends I want to do: Always | 2 | 1

55. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the Cocci Positive mITT Population
Description: as for outcome 43
Time Frame: Visit 4 (Day 42-46)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 0 | 0
  Trouble doing regular leisure activities w others: Sometimes | 1 | 0
  Trouble doing regular leisure activities w others: Usually | 0 | 0
  Trouble doing regular leisure activities w others: Always | 3 | 2
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 0 | 0
  Trouble doing family activities I want to do: Sometimes | 1 | 0
  Trouble doing family activities I want to do: Usually | 0 | 0
  Trouble doing family activities I want to do: Always | 3 | 2
  Trouble doing usual work (incl work at home): Never | 0 | 0
  Trouble doing usual work (incl work at home): Rarely | 1 | 0
  Trouble doing usual work (incl work at home): Sometimes | 0 | 0
  Trouble doing usual work (incl work at home): Usually | 0 | 1
  Trouble doing usual work (incl work at home): Always | 3 | 1
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 0 | 0
  Trouble doing activities with friends I want to do: Sometimes | 1 | 0
  Trouble doing activities with friends I want to do: Usually | 0 | 0
  Trouble doing activities with friends I want to do: Always | 3 | 2

56. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the Cocci Positive mITT Population
Description: as for outcome 43
Time Frame: Visit 6 (Day 83-97)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 0 | 0
  Trouble doing regular leisure activities w others: Sometimes | 1 | 0
  Trouble doing regular leisure activities w others: Usually | 0 | 0
  Trouble doing regular leisure activities w others: Always | 3 | 1
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 0 | 0
  Trouble doing family activities I want to do: Sometimes | 1 | 0
  Trouble doing family activities I want to do: Usually | 0 | 0
  Trouble doing family activities I want to do: Always | 3 | 1
  Trouble doing usual work (incl work at home): Never | 1 | 0
  Trouble doing usual work (incl work at home): Rarely | 0 | 0
  Trouble doing usual work (incl work at home): Sometimes | 0 | 0
  Trouble doing usual work (incl work at home): Usually | 0 | 0
  Trouble doing usual work (incl work at home): Always | 3 | 1
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 0 | 0
  Trouble doing activities with friends I want to do: Sometimes | 1 | 0
  Trouble doing activities with friends I want to do: Usually | 0 | 0
  Trouble doing activities with friends I want to do: Always | 3 | 1

57. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the Cocci Positive mITT Population
Description: as for outcome 43
Time Frame: Visit 7 (Day 173-187)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 1 | 0
  Trouble doing regular leisure activities w others: Sometimes | 0 | 0
  Trouble doing regular leisure activities w others: Usually | 0 | 0
  Trouble doing regular leisure activities w others: Always | 3 | 1
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 0 | 0
  Trouble doing family activities I want to do: Sometimes | 0 | 0
  Trouble doing family activities I want to do: Usually | 1 | 0
  Trouble doing family activities I want to do: Always | 3 | 1
  Trouble doing usual work (incl work at home): Never | 0 | 0
  Trouble doing usual work (incl work at home): Rarely | 0 | 0
  Trouble doing usual work (incl work at home): Sometimes | 1 | 0
  Trouble doing usual work (incl work at home): Usually | 0 | 0
  Trouble doing usual work (incl work at home): Always | 3 | 1
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 1 | 0
  Trouble doing activities with friends I want to do: Sometimes | 0 | 0
  Trouble doing activities with friends I want to do: Usually | 0 | 0
  Trouble doing activities with friends I want to do: Always | 3 | 1

58. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the All Randomized Per Protocol Population
Description: as for outcome 43
Time Frame: Visit 2 (Day 20-23)
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 25 | 29
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 1
  Trouble doing regular leisure activities w others: Rarely | 1 | 4
  Trouble doing regular leisure activities w others: Sometimes | 7 | 8
  Trouble doing regular leisure activities w others: Usually | 3 | 7
  Trouble doing regular leisure activities w others: Always | 14 | 9
  Trouble doing family activities I want to do: Never | 0 | 1
  Trouble doing family activities I want to do: Rarely | 2 | 4
  Trouble doing family activities I want to do: Sometimes | 4 | 7
  Trouble doing family activities I want to do: Usually | 5 | 6
  Trouble doing family activities I want to do: Always | 14 | 11
  Trouble doing usual work (incl work at home): Never | 0 | 1
  Trouble doing usual work (incl work at home): Rarely | 5 | 4
  Trouble doing usual work (incl work at home): Sometimes | 5 | 9
  Trouble doing usual work (incl work at home): Usually | 4 | 6
  Trouble doing usual work (incl work at home): Always | 11 | 9
  Trouble doing activities with friends I want to do: Never | 0 | 2
  Trouble doing activities with friends I want to do: Rarely | 3 | 2
  Trouble doing activities with friends I want to do: Sometimes | 5 | 10
  Trouble doing activities with friends I want to do: Usually | 4 | 7
  Trouble doing activities with friends I want to do: Always | 13 | 8

59. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the All Randomized Per Protocol Population
Description: as for outcome 43
Time Frame: Visit 3 (Day 27-30)
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 24 | 25
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 3 | 1
  Trouble doing regular leisure activities w others: Sometimes | 5 | 6
  Trouble doing regular leisure activities w others: Usually | 4 | 13
  Trouble doing regular leisure activities w others: Always | 12 | 5
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 2 | 1
  Trouble doing family activities I want to do: Sometimes | 5 | 9
  Trouble doing family activities I want to do: Usually | 4 | 10
  Trouble doing family activities I want to do: Always | 13 | 5
  Trouble doing usual work (incl work at home): Never | 0 | 0
  Trouble doing usual work (incl work at home): Rarely | 4 | 3
  Trouble doing usual work (incl work at home): Sometimes | 4 | 8
  Trouble doing usual work (incl work at home): Usually | 4 | 9
  Trouble doing usual work (incl work at home): Always | 12 | 5
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 2 | 3
  Trouble doing activities with friends I want to do: Sometimes | 5 | 6
  Trouble doing activities with friends I want to do: Usually | 5 | 9
  Trouble doing activities with friends I want to do: Always | 12 | 7

60. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the All Randomized Per Protocol Population
Description: as for outcome 43
Time Frame: Visit 4 (Day 42-46)
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 23 | 24
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 1 | 4
  Trouble doing regular leisure activities w others: Sometimes | 5 | 5
  Trouble doing regular leisure activities w others: Usually | 4 | 8
  Trouble doing regular leisure activities w others: Always | 13 | 7
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 2 | 4
  Trouble doing family activities I want to do: Sometimes | 4 | 4
  Trouble doing family activities I want to do: Usually | 2 | 6
  Trouble doing family activities I want to do: Always | 15 | 10
  Trouble doing usual work (incl work at home): Never | 1 | 0
  Trouble doing usual work (incl work at home): Rarely | 1 | 4
  Trouble doing usual work (incl work at home): Sometimes | 4 | 3
  Trouble doing usual work (incl work at home): Usually | 4 | 9
  Trouble doing usual work (incl work at home): Always | 13 | 8
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 2 | 4
  Trouble doing activities with friends I want to do: Sometimes | 4 | 5
  Trouble doing activities with friends I want to do: Usually | 4 | 4
  Trouble doing activities with friends I want to do: Always | 13 | 11

61. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the All Randomized Per Protocol Population
Description: as for outcome 43
Time Frame: Visit 6 (Day 83-97)
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 0 | 0
  Trouble doing regular leisure activities w others: Sometimes | 1 | 0
  Trouble doing regular leisure activities w others: Usually | 0 | 0
  Trouble doing regular leisure activities w others: Always | 3 | 1
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 0 | 0
  Trouble doing family activities I want to do: Sometimes | 1 | 0
  Trouble doing family activities I want to do: Usually | 0 | 0
  Trouble doing family activities I want to do: Always | 3 | 1
  Trouble doing usual work (incl work at home): Never | 1 | 0
  Trouble doing usual work (incl work at home): Rarely | 0 | 0
  Trouble doing usual work (incl work at home): Sometimes | 0 | 0
  Trouble doing usual work (incl work at home): Usually | 0 | 0
  Trouble doing usual work (incl work at home): Always | 3 | 1
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 0 | 0
  Trouble doing activities with friends I want to do: Sometimes | 1 | 0
  Trouble doing activities with friends I want to do: Usually | 0 | 0
  Trouble doing activities with friends I want to do: Always | 3 | 1

62. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the All Randomized Per Protocol Population
Description: as for outcome 43
Time Frame: Visit 7 (Day 173-187)
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 1 | 0
  Trouble doing regular leisure activities w others: Sometimes | 0 | 0
  Trouble doing regular leisure activities w others: Usually | 0 | 0
  Trouble doing regular leisure activities w others: Always | 3 | 1
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 0 | 0
  Trouble doing family activities I want to do: Sometimes | 0 | 0
  Trouble doing family activities I want to do: Usually | 1 | 0
  Trouble doing family activities I want to do: Always | 3 | 1
  Trouble doing usual work (incl work at home): Never | 0 | 0
  Trouble doing usual work (incl work at home): Rarely | 0 | 0
  Trouble doing usual work (incl work at home): Sometimes | 1 | 0
  Trouble doing usual work (incl work at home): Usually | 0 | 0
  Trouble doing usual work (incl work at home): Always | 3 | 1
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 1 | 0
  Trouble doing activities with friends I want to do: Sometimes | 0 | 0
  Trouble doing activities with friends I want to do: Usually | 0 | 0
  Trouble doing activities with friends I want to do: Always | 3 | 1

63. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the All Randomized mITT Population
Description: as for outcome 43
Time Frame: Visit 2 (Day 20-23)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 27 | 35
Participants
  Trouble doing regular leisure activities w others: Never | 1 | 3
  Trouble doing regular leisure activities w others: Rarely | 1 | 4
  Trouble doing regular leisure activities w others: Sometimes | 7 | 8
  Trouble doing regular leisure activities w others: Usually | 3 | 7
  Trouble doing regular leisure activities w others: Always | 15 | 13
  Trouble doing family activities I want to do: Never | 0 | 3
  Trouble doing family activities I want to do: Rarely | 3 | 4
  Trouble doing family activities I want to do: Sometimes | 4 | 7
  Trouble doing family activities I want to do: Usually | 5 | 6
  Trouble doing family activities I want to do: Always | 15 | 15
  Trouble doing usual work (incl work at home): Never | 0 | 3
  Trouble doing usual work (incl work at home): Rarely | 5 | 4
  Trouble doing usual work (incl work at home): Sometimes | 7 | 9
  Trouble doing usual work (incl work at home): Usually | 4 | 6
  Trouble doing usual work (incl work at home): Always | 11 | 13
  Trouble doing activities with friends I want to do: Never | 1 | 4
  Trouble doing activities with friends I want to do: Rarely | 3 | 2
  Trouble doing activities with friends I want to do: Sometimes | 5 | 10
  Trouble doing activities with friends I want to do: Usually | 4 | 7
  Trouble doing activities with friends I want to do: Always | 14 | 12

64. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the All Randomized mITT Population
Description: as for outcome 43
Time Frame: Visit 3 (Day 27-30)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 26 | 31
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 3 | 1
  Trouble doing regular leisure activities w others: Sometimes | 6 | 8
  Trouble doing regular leisure activities w others: Usually | 4 | 13
  Trouble doing regular leisure activities w others: Always | 13 | 9
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 2 | 1
  Trouble doing family activities I want to do: Sometimes | 6 | 11
  Trouble doing family activities I want to do: Usually | 4 | 10
  Trouble doing family activities I want to do: Always | 14 | 9
  Trouble doing usual work (incl work at home): Never | 0 | 0
  Trouble doing usual work (incl work at home): Rarely | 4 | 3
  Trouble doing usual work (incl work at home): Sometimes | 5 | 10
  Trouble doing usual work (incl work at home): Usually | 4 | 10
  Trouble doing usual work (incl work at home): Always | 13 | 8
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 2 | 3
  Trouble doing activities with friends I want to do: Sometimes | 6 | 7
  Trouble doing activities with friends I want to do: Usually | 5 | 10
  Trouble doing activities with friends I want to do: Always | 13 | 11

65. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the All Randomized mITT Population
Description: as for outcome 43
Time Frame: Visit 4 (Day 42-46)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 25 | 30
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 1 | 4
  Trouble doing regular leisure activities w others: Sometimes | 6 | 6
  Trouble doing regular leisure activities w others: Usually | 4 | 8
  Trouble doing regular leisure activities w others: Always | 14 | 12
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 2 | 4
  Trouble doing family activities I want to do: Sometimes | 5 | 5
  Trouble doing family activities I want to do: Usually | 2 | 6
  Trouble doing family activities I want to do: Always | 16 | 15
  Trouble doing usual work (incl work at home): Never | 1 | 0
  Trouble doing usual work (incl work at home): Rarely | 1 | 4
  Trouble doing usual work (incl work at home): Sometimes | 5 | 4
  Trouble doing usual work (incl work at home): Usually | 4 | 11
  Trouble doing usual work (incl work at home): Always | 14 | 11
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 2 | 5
  Trouble doing activities with friends I want to do: Sometimes | 5 | 5
  Trouble doing activities with friends I want to do: Usually | 4 | 4
  Trouble doing activities with friends I want to do: Always | 14 | 16

66. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the All Randomized mITT Population
Description: as for outcome 43
Time Frame: Visit 6 (Day 83-97)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 0 | 0
  Trouble doing regular leisure activities w others: Sometimes | 1 | 0
  Trouble doing regular leisure activities w others: Usually | 0 | 0
  Trouble doing regular leisure activities w others: Always | 3 | 1
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 0 | 0
  Trouble doing family activities I want to do: Sometimes | 1 | 0
  Trouble doing family activities I want to do: Usually | 0 | 0
  Trouble doing family activities I want to do: Always | 3 | 1
  Trouble doing usual work (incl work at home): Never | 1 | 0
  Trouble doing usual work (incl work at home): Rarely | 0 | 0
  Trouble doing usual work (incl work at home): Sometimes | 0 | 0
  Trouble doing usual work (incl work at home): Usually | 0 | 0
  Trouble doing usual work (incl work at home): Always | 3 | 1
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 0 | 0
  Trouble doing activities with friends I want to do: Sometimes | 1 | 0
  Trouble doing activities with friends I want to do: Usually | 0 | 0
  Trouble doing activities with friends I want to do: Always | 3 | 1

67. Secondary Outcome: Number of Participants Responding to the Individual Items of the PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a in the All Randomized mITT Population
Description: as for outcome 43
Time Frame: Visit 7 (Day 173-187)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
Participants
  Trouble doing regular leisure activities w others: Never | 0 | 0
  Trouble doing regular leisure activities w others: Rarely | 1 | 0
  Trouble doing regular leisure activities w others: Sometimes | 0 | 0
  Trouble doing regular leisure activities w others: Usually | 0 | 0
  Trouble doing regular leisure activities w others: Always | 3 | 1
  Trouble doing family activities I want to do: Never | 0 | 0
  Trouble doing family activities I want to do: Rarely | 0 | 0
  Trouble doing family activities I want to do: Sometimes | 0 | 0
  Trouble doing family activities I want to do: Usually | 1 | 0
  Trouble doing family activities I want to do: Always | 3 | 1
  Trouble doing usual work (incl work at home): Never | 0 | 0
  Trouble doing usual work (incl work at home): Rarely | 0 | 0
  Trouble doing usual work (incl work at home): Sometimes | 1 | 0
  Trouble doing usual work (incl work at home): Usually | 0 | 0
  Trouble doing usual work (incl work at home): Always | 3 | 1
  Trouble doing activities with friends I want to do: Never | 0 | 0
  Trouble doing activities with friends I want to do: Rarely | 1 | 0
  Trouble doing activities with friends I want to do: Sometimes | 0 | 0
  Trouble doing activities with friends I want to do: Usually | 0 | 0
  Trouble doing activities with friends I want to do: Always | 3 | 1

68. Secondary Outcome: Incidence Rate of All-cause Mortality
Description: Mortality information was obtained through medical records or next of kin.
Time Frame: Day 1 through Day 43
Population: The population includes all participants who took at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 25 | 30
participants | 0 | 0

69. Secondary Outcome: The Proportion of Participants Who Achieve a Clinical Response, Defined as at Least a 50% Reduction in Composite FLEET CAP Score From Baseline, in All Randomized Participants, Regardless of Coccidioidomycosis Status or Adherence to Study Drug
Description: as for outcome 1
Time Frame: Visit 2 (Day 20-23)
Population: Intent-to-Treat (ITT) population - This efficacy analysis population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 27 | 35
Participants | 20 | 22

70. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, ITT Population
Description: The SF-12v2 uses 12 questions to measure functional health and well-being from the study participant's perspective across eight domains: physical functioning, role, bodily pain, general health perceptions, vitality, social functioning, emotional role, and mental health. Mental and physical composite scores (MCS & PCS) are computed using the scores of twelve questions and range from 0 to 100, where a higher score indicates better health.
Time Frame: Day 1
Population: The Intent-to-Treat (ITT) population includes all randomized participants with data at the time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 32 | 39
score on a scale
  MCS | 48.2 (10.1) | 49.0 (10.2)
  PCS | 38.6 (11.1) | 39.7 (9.8)

71. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, ITT Population
Description: as for outcome 70
Time Frame: Day 22
Population: The Intent-to-Treat (ITT) population includes all randomized participants with data at the time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 27 | 35
score on a scale
  MCS | 51.4 (10.0) | 49.4 (10.7)
  PCS | 45.4 (11.2) | 44.2 (12.0)

72. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, ITT Population
Description: as for outcome 70
Time Frame: Day 29
Population: The Intent-to-Treat (ITT) population includes all randomized participants with data at the time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 26 | 31
score on a scale
  MCS | 49.5 (10.6) | 50.6 (9.9)
  PCS | 47.9 (10.5) | 46.2 (11.5)

73. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, ITT Population
Description: as for outcome 70
Time Frame: Day 43
Population: The Intent-to-Treat (ITT) population includes all randomized participants with data at the time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 24 | 30
score on a scale
  MCS | 52.4 (10.0) | 51.3 (8.7)
  PCS | 50.1 (8.9) | 46.2 (11.2)

74. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, ITT Population
Description: as for outcome 70
Time Frame: Day 90
Population: The Intent-to-Treat (ITT) population includes all randomized participants with data at the time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
score on a scale
  MCS | 51.5 (13.1) | 49.5
  PCS | 52.9 (9.0) | 55.5

75. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, ITT Population
Description: as for outcome 70
Time Frame: Day 180
Population: The Intent-to-Treat (ITT) population includes all randomized participants with data at the time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
score on a scale
  MCS | 55.3 (9.8) | 61.1
  PCS | 46.9 (9.1) | 57.7

76. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci Positive PP Population
Description: as for outcome 70
Time Frame: Day 1
Population: The cocci-positive per-protocol population includes randomized participants who met the case definition of cocci pneumonia, were adherent with the intervention and had coccidioidal serology data available at the Day 1 and 22 visits. To be considered adherent at the Day 22 visit, the subject needed to take >=80% of their expected pills.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  MCS | 52.0 (6.3) | 37.1 (8.3)
  PCS | 46.2 (15.4) | 45.3 (1.9)

77. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci Positive PP Population
Description: as for outcome 70
Time Frame: Day 22
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  MCS | 51.6 (8.3) | 43.7 (9.6)
  PCS | 49.6 (12.3) | 60.1 (1.5)

78. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci Positive PP Population
Description: as for outcome 70
Time Frame: Day 29
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  MCS | 54.0 (11.3) | 43.9 (24.3)
  PCS | 51.6 (11.0) | 60.1 (3.4)

79. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci Positive PP Population
Description: as for outcome 70
Time Frame: Day 43
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  MCS | 53.6 (12.2) | 50.2 (15.5)
  PCS | 53.6 (7.0) | 58.9 (1.7)

80. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci Positive PP Population
Description: as for outcome 70
Time Frame: Day 90
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
score on a scale
  MCS | 51.5 (13.1) | 49.5
  PCS | 52.9 (9.0) | 55.5

81. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci Positive PP Population
Description: as for outcome 70
Time Frame: Day 180
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
score on a scale
  MCS | 55.3 (9.8) | 61.1
  PCS | 46.9 (9.1) | 57.7

82. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci Positive mITT Population
Description: as for outcome 70
Time Frame: Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 4
score on a scale
  MCS | 52.0 (6.3) | 39.0 (12.3)
  PCS | 46.2 (15.4) | 42.2 (10.5)

83. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci Positive mITT Population
Description: as for outcome 70
Time Frame: Day 22
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 3
score on a scale
  MCS | 51.6 (8.3) | 40.6 (8.7)
  PCS | 49.6 (12.3) | 47.4 (22.1)

84. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci Positive mITT Population
Description: as for outcome 70
Time Frame: Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  MCS | 54.0 (11.3) | 43.9 (24.3)
  PCS | 51.6 (11.0) | 60.1 (3.4)

85. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci Positive mITT Population
Description: as for outcome 70
Time Frame: Day 43
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  MCS | 53.6 (12.2) | 50.2 (15.5)
  PCS | 53.6 (7.0) | 58.9 (1.7)

86. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci Positive mITT Population
Description: as for outcome 70
Time Frame: Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
score on a scale
  MCS | 51.5 (13.1) | 49.5
  PCS | 52.9 (9.0) | 55.5

87. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci Positive mITT Population
Description: as for outcome 70
Time Frame: Day 180
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
score on a scale
  MCS | 55.3 (9.8) | 61.1
  PCS | 46.9 (9.1) | 57.7

88. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized PP Population
Description: as for outcome 70
Time Frame: Day 1
Population: The All-Randomized PP population includes all participants who took at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 24 | 29
score on a scale
  MCS | 49.1 (10.2) | 47.9 (9.5)
  PCS | 39.4 (11.6) | 39.6 (10.0)

89. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized PP Population
Description: as for outcome 70
Time Frame: Day 22
Population: The All-Randomized PP population includes all participants who took at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 25 | 29
score on a scale
  MCS | 51.7 (9.3) | 49.6 (10.8)
  PCS | 45.9 (11.3) | 43.2 (11.4)

90. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized PP Population
Description: as for outcome 70
Time Frame: Day 29
Population: The All-Randomized PP population includes all participants who took at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 24 | 25
score on a scale
  MCS | 50.5 (10.2) | 50.8 (10.3)
  PCS | 48.3 (10.7) | 45.3 (11.9)

91. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized PP Population
Description: as for outcome 70
Time Frame: Day 43
Population: The All-Randomized PP population includes all participants who took at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 22 | 24
score on a scale
  MCS | 53.3 (10.0) | 49.8 (9.0)
  PCS | 50.5 (9.1) | 46.0 (11.0)

92. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized PP Population
Description: as for outcome 70
Time Frame: Day 90
Population: The All-Randomized PP population includes all participants who took at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
score on a scale
  MCS | 51.5 (13.1) | 49.5
  PCS | 52.9 (9.0) | 55.5

93. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized PP Population
Description: as for outcome 70
Time Frame: Day 180
Population: The All-Randomized PP population includes all participants who took at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
score on a scale
  MCS | 55.3 (9.8) | 61.1
  PCS | 46.9 (9.1) | 57.7

94. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized mITT Population
Description: as for outcome 70
Time Frame: Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 32 | 39
score on a scale
  MCS | 48.2 (10.1) | 49.0 (10.2)
  PCS | 38.6 (11.1) | 39.7 (9.8)

95. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized mITT Population
Description: as for outcome 70
Time Frame: Day 22
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 27 | 35
score on a scale
  MCS | 51.4 (10.0) | 49.4 (10.7)
  PCS | 45.4 (11.2) | 44.2 (12.0)

96. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized mITT Population
Description: as for outcome 70
Time Frame: Day 29
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 26 | 31
score on a scale
  MCS | 49.5 (10.6) | 50.6 (9.9)
  PCS | 47.9 (10.5) | 46.2 (11.5)

97. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized mITT Population
Description: as for outcome 70
Time Frame: Day 43
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 24 | 30
score on a scale
  MCS | 52.4 (10.0) | 51.3 (8.7)
  PCS | 50.1 (8.9) | 46.2 (11.2)

98. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized mITT Population
Description: as for outcome 70
Time Frame: Day 90
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
score on a scale
  MCS | 51.5 (13.1) | 49.5
  PCS | 52.9 (9.0) | 55.5

99. Secondary Outcome: The Mean for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized mITT Population
Description: as for outcome 70
Time Frame: Day 180
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
score on a scale
  MCS | 55.3 (9.8) | 61.1
  PCS | 46.9 (9.1) | 57.7

100. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, ITT Population
Description: as for outcome 70
Time Frame: Day 1
Population: The Intent-to-Treat (ITT) population includes all randomized participants with data at the time point.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 32 | 39
score on a scale
  MCS | 50.0 [41.1 to 56.4] | 49.6 [42.0 to 56.1]
  PCS | 39.1 [30.1 to 45.2] | 39.1 [31.9 to 46.7]

101. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, ITT Population
Description: as for outcome 70
Time Frame: Day 22
Population: The Intent-to-Treat (ITT) population includes all randomized participants with data at the time point.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 27 | 35
score on a scale
  MCS | 54.9 [44.5 to 59.1] | 50.5 [43.1 to 59.1]
  PCS | 46.5 [35.5 to 55.7] | 46.0 [33.4 to 56.0]

102. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, ITT Population
Description: as for outcome 70
Time Frame: Day 29
Population: The Intent-to-Treat (ITT) population includes all randomized participants with data at the time point.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 26 | 31
score on a scale
  MCS | 54.5 [40.2 to 57.8] | 52.9 [43.1 to 58.2]
  PCS | 52.5 [39.3 to 57.2] | 47.5 [36.8 to 57.2]

103. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, ITT Population
Description: as for outcome 70
Time Frame: Day 43
Population: The Intent-to-Treat (ITT) population includes all randomized participants with data at the time point.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 24 | 30
score on a scale
  MCS | 56.4 [43.1 to 60.2] | 54.1 [46.6 to 59.0]
  PCS | 53.5 [44.8 to 56.7] | 48.6 [41.2 to 53.8]

104. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, ITT Population
Description: as for outcome 70
Time Frame: Day 90
Population: The Intent-to-Treat (ITT) population includes all randomized participants with data at the time point.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
score on a scale
  MCS | 56.4 [44.3 to 58.8] | 49.5 [49.5 to 49.5]
  PCS | 57.2 [48.3 to 57.5] | 55.5 [55.5 to 55.5]

105. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, ITT Population
Description: as for outcome 70
Time Frame: Day 180
Population: The Intent-to-Treat (ITT) population includes all randomized participants with data at the time point.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
score on a scale
  MCS | 59.2 [49.2 to 61.5] | 61.1 [61.1 to 61.1]
  PCS | 50.9 [41.7 to 52.1] | 57.7 [57.7 to 57.7]

106. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci-positive Per-protocol Population
Description: as for outcome 70
Time Frame: Day 1
Population: as for outcome 26
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  MCS | 52.7 [46.8 to 57.2] | 37.1 [31.3 to 43.0]
  PCS | 51.2 [35.0 to 57.4] | 45.3 [43.9 to 46.7]

107. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci-positive Per-protocol Population
Description: as for outcome 70
Time Frame: Day 22
Population: as for outcome 26
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  MCS | 54.5 [46.7 to 56.5] | 43.7 [36.9 to 50.5]
  PCS | 53.5 [42.2 to 57.0] | 60.1 [59.0 to 61.1]

108. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci-positive Per-protocol Population
Description: as for outcome 70
Time Frame: Day 29
Population: as for outcome 26
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  MCS | 58.8 [46.9 to 61.2] | 43.9 [26.8 to 61.1]
  PCS | 56.7 [45.6 to 57.5] | 60.1 [57.7 to 62.5]

109. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci-positive Per-protocol Population
Description: as for outcome 70
Time Frame: Day 43
Population: as for outcome 26
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  MCS | 58.8 [46.0 to 61.2] | 50.2 [39.2 to 61.1]
  PCS | 56.7 [49.7 to 57.5] | 58.9 [57.7 to 60.1]

110. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci-positive Per-protocol Population
Description: as for outcome 70
Time Frame: Day 90
Population: as for outcome 26
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
score on a scale
  MCS | 56.4 [44.3 to 58.8] | 49.5 [49.5 to 49.5]
  PCS | 57.2 [48.3 to 57.5] | 55.5 [55.5 to 55.5]

111. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci-positive Per-protocol Population
Description: as for outcome 70
Time Frame: Day 180
Population: as for outcome 26
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
score on a scale
  MCS | 59.2 [49.2 to 61.5] | 61.1 [61.1 to 61.1]
  PCS | 50.9 [41.7 to 52.1] | 57.7 [57.7 to 57.7]

112. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci Positive Modified Intent-to-Treat Population
Description: as for outcome 70
Time Frame: Day 1
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 4
score on a scale
  MCS | 52.7 [46.8 to 57.2] | 37.1 [29.3 to 48.8]
  PCS | 51.2 [35.0 to 57.4] | 45.3 [35.6 to 48.9]

113. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci Positive Modified Intent-to-Treat Population
Description: as for outcome 70
Time Frame: Day 22
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 3
score on a scale
  MCS | 54.5 [46.7 to 56.5] | 36.9 [34.4 to 50.5]
  PCS | 53.5 [42.2 to 57.0] | 59.0 [21.9 to 61.1]

114. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci Positive Modified Intent-to-Treat Population
Description: as for outcome 70
Time Frame: Day 29
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  MCS | 58.8 [46.9 to 61.2] | 43.9 [26.8 to 61.1]
  PCS | 56.7 [45.6 to 57.5] | 60.1 [57.7 to 62.5]

115. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci Positive Modified Intent-to-Treat Population
Description: as for outcome 70
Time Frame: Day 43
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  MCS | 58.8 [46.0 to 61.2] | 50.2 [39.2 to 61.1]
  PCS | 56.7 [49.7 to 57.5] | 58.9 [57.7 to 60.1]

116. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci Positive Modified Intent-to-Treat Population
Description: as for outcome 70
Time Frame: Day 90
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
score on a scale
  MCS | 56.4 [44.3 to 58.8] | 49.5 [49.5 to 49.5]
  PCS | 57.2 [48.3 to 57.5] | 55.5 [55.5 to 55.5]

117. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, Cocci Positive Modified Intent-to-Treat Population
Description: as for outcome 70
Time Frame: Day 180
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
score on a scale
  MCS | 59.2 [49.2 to 61.5] | 61.1 [61.1 to 61.1]
  PCS | 50.9 [41.7 to 52.1] | 57.7 [57.7 to 57.7]

118. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized PP Population
Description: as for outcome 70
Time Frame: Day 1
Population: The All-Randomized PP population includes all participants who took at least one dose of study medication.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 24 | 29
score on a scale
  MCS | 51.1 [44.4 to 56.4] | 47.9 [40.7 to 54.9]
  PCS | 39.7 [31.1 to 46.5] | 39.2 [31.9 to 46.1]

119. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized PP Population
Description: as for outcome 70
Time Frame: Day 22
Population: The All-Randomized PP population includes all participants who took at least one dose of study medication.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 25 | 29
score on a scale
  MCS | 54.9 [44.7 to 58.5] | 50.5 [43.1 to 59.1]
  PCS | 48.3 [36.3 to 55.7] | 45.3 [33.4 to 53.2]

120. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized PP Population
Description: as for outcome 70
Time Frame: Day 29
Population: The All-Randomized PP population includes all participants who took at least one dose of study medication.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 24 | 25
score on a scale
  MCS | 55.6 [42.9 to 58.3] | 53.3 [44.2 to 58.2]
  PCS | 52.9 [40.0 to 57.2] | 46.9 [36.8 to 54.8]

121. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized PP Population
Description: as for outcome 70
Time Frame: Day 43
Population: The All-Randomized PP population includes all participants who took at least one dose of study medication.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 22 | 24
score on a scale
  MCS | 57.2 [51.7 to 61.1] | 49.6 [43.3 to 58.4]
  PCS | 54.0 [46.3 to 57.2] | 48.2 [38.5 to 53.6]

122. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized PP Population
Description: as for outcome 70
Time Frame: Day 90
Population: The All-Randomized PP population includes all participants who took at least one dose of study medication.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
score on a scale
  MCS | 56.4 [44.3 to 58.8] | 49.5 [49.5 to 49.5]
  PCS | 57.2 [48.3 to 57.5] | 55.5 [55.5 to 55.5]

123. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized PP Population
Description: as for outcome 70
Time Frame: Day 180
Population: The All-Randomized PP population includes all participants who took at least one dose of study medication.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
score on a scale
  MCS | 59.2 [49.2 to 61.5] | 61.1 [61.1 to 61.1]
  PCS | 50.9 [41.7 to 52.1] | 57.7 [57.7 to 57.7]

124. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized mITT Population
Description: as for outcome 70
Time Frame: Day 1
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 32 | 39
score on a scale
  MCS | 50.0 [41.1 to 56.4] | 49.6 [42.0 to 56.1]
  PCS | 39.1 [30.1 to 45.2] | 39.1 [31.9 to 46.7]

125. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized mITT Population
Description: as for outcome 70
Time Frame: Day 22
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 27 | 35
score on a scale
  MCS | 54.9 [44.5 to 59.1] | 50.5 [43.1 to 59.1]
  PCS | 46.5 [35.5 to 55.7] | 46.0 [33.4 to 56.0]

126. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized mITT Population
Description: as for outcome 70
Time Frame: Day 29
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 26 | 31
score on a scale
  MCS | 54.5 [40.2 to 57.8] | 52.9 [43.1 to 58.2]
  PCS | 52.5 [39.3 to 57.2] | 47.5 [36.8 to 57.2]

127. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized mITT Population
Description: as for outcome 70
Time Frame: Day 43
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 24 | 30
score on a scale
  MCS | 56.4 [43.1 to 60.2] | 54.1 [46.6 to 59.0]
  PCS | 53.5 [44.8 to 56.7] | 48.6 [41.2 to 53.8]

128. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized mITT Population
Description: as for outcome 70
Time Frame: Day 90
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
score on a scale
  MCS | 56.4 [44.3 to 58.8] | 49.5 [49.5 to 49.5]
  PCS | 57.2 [48.3 to 57.5] | 55.5 [55.5 to 55.5]

129. Secondary Outcome: The Median for the Mental Component Summary (MCS) and the Physical Component Summary (PCS) Scores of the SF-12v2 Instrument, All Randomized mITT Population
Description: as for outcome 70
Time Frame: Day 180
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 4 | 1
score on a scale
  MCS | 59.2 [49.2 to 61.5] | 61.1 [61.1 to 61.1]
  PCS | 50.9 [41.7 to 52.1] | 57.7 [57.7 to 57.7]

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from the time of enrollment until completion of study.
Description: The safety data collection was targeted to only collect Suspected Unexpected Serious Adverse Reactions (SUSARs) and congenital anomalies/birth defects. Non-serious adverse events were not collected.
Arm/Group | Fluconazole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/39
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study terminated early due to low enrollment rates. When the study was stopped, 72 of a planned 1000 participants were enrolled and randomized; therefore, formal comparisons of the endpoints are not included.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/74/NCT02663674/Prot_SAP_000.pdf